CLINICAL TRIAL: NCT05010954
Title: A Multi-center, Randomized, Double-blind, Active-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of LXI-15028 Compared to Lansoprazole in the Treatment of Duodenal Ulcer in Chinese Patients for up to 6 Weeks
Brief Title: Efficacy and Safety of LXI-15028 Comparing With Lansoprazole in the Treatment of Duodenal Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC821604
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Duodenal Ulcer
MeSH Terms: conditions — Duodenal Ulcer | interventions — Population Groups; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LXI-15028 50mg group(n=200) (Experimental)
  Interventions: Drug: LXI-15028 50mg group
- Lansoprazole 30mg group (n=200) (Active Comparator)
  Interventions: Drug: Lansoprazole 30mg group

INTERVENTIONS:
Drug: LXI-15028 50mg group — The investigational products are administrated orally, once in the morning every day, and each dose includes 2 tablets of investigational products (LXI-15028 50mg active agent + Lansoprazole 30mg matching placebo). If the investigational product is not taken in the morning, subjects can take it before 6:00 p.m. on the same day. The duration of treatment is 4 or 6 weeks
  Arms: LXI-15028 50mg group(n=200)
Drug: Lansoprazole 30mg group — The investigational products are administrated orally, once in the morning every day, and each dose includes 2 tablets of investigational products ( LXI-15028 50mg matching placebo + Lansoprazole 30mg active agent ). If the investigational product is not taken in the morning, subjects can take it before 6:00 p.m. on the same day. The duration of treatment is 4 or 6 weeks.
  Arms: Lansoprazole 30mg group (n=200)

SUMMARY:
This is a multi-center, randomized, double-blind, double-dummy, parallel-group, active-controlled Phase III clinical study to evaluate the efficacy and safety of LXI-15028 50mg comparing with Lansoprazole 30 mg after the treatment of duodenal ulcer in Chinese patients for up to 6 weeks.

DETAILED DESCRIPTION:
Screening-eligible subjects will be randomized into LXI-15028 50 mg group or Lansoprazole 30 mg group at Visit 1 at the ratio of 1:1 and receive study treatment continuously for 4 or 6 weeks.Subjects will take the first dose of the investigational drug on the morning of the randomization day or on the next morning of the randomization day, and start to complete the subject's diary from the day of study treatment initiation(Day 1). After 4 weeks treatment, subjects will return to the study institution for Visit 3. For the subjects who achieve endoscopic healing at Visit 3,the study treatment will be terminated.The subjects who fail to achieve endoscopic healing at Visit 3 will receive newly dispensed investigational products for another 2 weeks' treatment and then complete Visit 4.All subjects will receive telephone follow-up (Visit 5) on Day 28 ± 3 after the last dose of the investigational products.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who volunteers to sign the written informed consent form approved by the Ethics Committee and agrees to participate in this study prior to the initiation of any study procedures.
2. Subject who is able to understand and follow the protocol requirements and agrees to participate in all the study visits.
3. Male or female subjects with age ≥18 years and ≤70 years.
4. Subject who is diagnosed as active DU (at least one ulcer, but not more than two ulcers, with the bigger one 0.3-2.0 cm in diameter) by upper gastrointestinal tract endoscopy in the same study institution within 14 days prior to the first dose of investigational drug and is staged as A1 or A2 by using the staging system of Sakita-Miwa.
5. Subject who agrees to use appropriate medical method for contraception during the course of the study (not including women in medically sterile state)

Exclusion Criteria:

1. Subject who had participated in any other clinical study of LXI-15028 previously, or had been treated with any P-CAB drug before.
2. Participation in other clinical study within 4 weeks prior to the first dose of study drug, except for the two following circumstances:

   1. The study which the subject is participating or participated in is a non-interventional study (e.g. observational study or questionnaire survey) and is judged by investigators to have no interference with the efficacy and safety evaluation in the present study;
   2. Subject had signed the informed consent form in that study, but withdrew from that study prior to the start of any treatment.
3. Subject who participates in the planning or conduct of this study.
4. Pregnant or lactating women.
5. Subject who is known to be allergic to the active ingredient or excipient of the investigational drug (including Lansoprazole).
6. Subject who is unable to undertake an upper gastrointestinal tract endoscopy.
7. Subject who is unable to complete the subject diary by his/her own.
8. Subject who has history of manic-depression, somatoform disorder, personality disorder, schizophrenia or other severe mental disorder.
9. Ulcers caused by endoscopic procedures, e.g. post endoscopic mucosal resection (EMR)/endoscopic submucosal dissection (ESD) ulcers.
10. Zollinger-Ellison syndrome.
11. History of malignant tumor within 5 years prior to screening (if the subject's basal cell carcinoma or cervical carcinoma in situ has been cured, he/she will be allowed to participate in this study).
12. Subject with history of upper GI surgery (except endoscopic surgery such as resection of benign polyp, etc.).
13. Subject who plans to be hospitalized for receiving selective surgery during the study.
14. Subject with uncontrolled and unstable hepatic, renal, cardiovascular, respiratory, endocrine, hematologic or central nervous system disease as judged by investigators.
15. Subject with history of chronic alcohol consumption [more than 14 units per week, each unit corresponds to 360 mL beer (ABV ≈ 5%) or 45 mL spirit (ABV ≈ 40%) or 150 mL wine (ABV ≈ 12%)] or drug abuse within 5 years prior to screening.
16. Subject whose upper gastrointestinal tract endoscopy shows GI bleeding (grade I, IIa or IIb per Forrest classification), esophageal stenosis, ulcerative stenosis, pyloric stenosis, gastroesophageal varices, Barrett's esophagus >3 cm (i.e., long-segment Barrett's esophagus, LSBE), gastroesophageal reflux disease, acute gastroduodenal mucosal lesion (AGDML), active gastric ulcer, refractory ulcer, ulcer perforation or suspected malignant disease.
17. Subject who has other severe GI diseases such as Crohn's disease, ulcerative colitis, etc.
18. Use of any PPI, anticholinergic drug, gastrin receptor antagonist, H2 receptor antagonist, prostaglandin, mucosal protective agent, prokinetic, antacid or any other therapeutic drugs for peptic ulcer within 14 days prior to the first dose of study drug.
19. Subject who has thrombotic disease (e.g., cerebral thrombosis, myocardial infarction, thrombophlebitis, etc.) or is currently on anticoagulant therapy.
20. Subject who needs to use nonsteroidal anti-inflammatory drugs (NSAIDs) continuously during the course of the study.
21. Use of any antipsychotic, antidepressant or anti-anxiety agent during screening.
22. Any of the following laboratory abnormalities at screening:

    * AST > Upper limit of normal (ULN);
    * ALT > ULN;
    * Total bilirubin > ULN;
    * Creatinine > 1.5 × ULN;
    * Platelet<lower limit of normal
    * Prothrombin time>1.5 × ULN
23. Subject who has clinically significant abnormality in electrocardiogram (ECG), including severe arrhythmia, multifocal premature ventricular contraction (PVC), Ⅱ or above atrioventricular block, etc.
24. Human immunodeficiency virus (HIV) antibody (+), hepatitis B virus (HBV) surface antigen (+) or hepatitis C virus (HCV) antibody (+) confirmed by tests.
25. Judged by the investigator, there are other conditions compromising the subject's eligibility for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Cumulative endoscopic healing rate | 4 or 6 weeks after receiving oral doses

SECONDARY OUTCOMES:
Endoscopic healing rate at Week 4 | 4 week after receiving oral doses
Symptom assessment based on subject diary | 4 or 6 weeks after receiving oral doses

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zong Y, Lan C, Li X, Chen W, Chen H, Liao A, Liu S, Hu C, Wu Y, Zhang S. Efficacy and safety of tegoprazan for duodenal ulcers in Chinese patients: a multicenter, randomized, double-blind, non-inferiority, phase III study. Curr Med Res Opin. 2024 Nov;40(11):1855-1862. doi: 10.1080/03007995.2024.2414090. Epub 2024 Oct 21. PMID 39378042